CLINICAL TRIAL: NCT00054145
Title: A Phase 2 Study Of Perifosine In Metastatic Or Advanced Breast Cancer
Brief Title: Perifosine in Treating Patients With Recurrent, Refractory, Locally Advanced, or Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: PMH-PHL-014; CDR0000269901 (Registry Identifier: PDQ (Physician Data Query)); NCI-5982
Record Dates: First submitted 2003-02-05; First posted 2003-02-06 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-07

CONDITIONS: Breast Cancer
Keywords: male breast cancer; recurrent breast cancer; stage IV breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — perifosine

INTERVENTIONS:
Drug: perifosine

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of perifosine in treating patients who have recurrent, refractory, locally advanced, or metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the objective tumor response rate in patients with recurrent or refractory, locally advanced or metastatic breast cancer treated with perifosine.
* Determine the toxicity of this drug in these patients.
* Determine the stable disease rate, time to disease progression, objective response duration, and duration of stable disease in patients treated with this drug.
* Correlate potential endpoints, including phosphorylated ERK, PKB, and SAPK, phosphorylated PKC alpha, beta, and gamma isoforms, p21 ^WAF1; and activated capase-3 in tumor biopsies, with clinical outcome in patients treated with this drug.

OUTLINE: This is an open-label, multicenter study.

Patients receive a loading dose of oral perifosine on days 1 and 2 and once daily on days 3-21 during course 1. Patients receive oral perifosine once daily on days 1-21 in each subsequent course. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients achieving a complete response (CR) may receive 2 additional courses beyond the CR.

PROJECTED ACCRUAL: A total of 18-35 patients will be accrued for this study within 6-12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed breast cancer

  * Recurrent or refractory, locally advanced or metastatic disease
* At least 1 unidimensionally measurable lesion

  * At least 20 mm by conventional techniques OR 10 mm by spiral CT scan
  * Previously irradiated lesions are not considered measurable unless they have demonstrated progression before study entry
  * No measurable disease limited to bone lesions
* No known brain metastases
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* 18 and over

Sex

* Male or female

Menopausal status

* Not specified

Performance status

* ECOG 0-2 OR
* Karnofsky 60-100%

Life expectancy

* More than 3 months

Hematopoietic

* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* No history of hemolytic disorder

Hepatic

* Bilirubin no greater than 1.25 times upper limit of normal (ULN)
* AST/ALT no greater than 2.5 times ULN (5 times ULN if liver metastases present)

Renal

* Creatinine normal OR
* Creatinine clearance at least 60 mL/min

Cardiovascular

* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* No evidence of cardiac dysfunction

Gastrointestinal

* No history of biliary flow obstruction
* No abnormalities of the gastrointestinal tract that would preclude study drug absorption
* No active peptic ulcer disease

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No ongoing or active infection
* No poorly controlled diabetes mellitus
* No other uncontrolled illness
* No prior allergic reactions to compounds of similar chemical or biological composition to perifosine
* No psychiatric illness or social situation that would preclude study compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No more than 2 prior lines of chemotherapy for advanced disease, excluding adjuvant chemotherapy
* Prior adjuvant chemotherapy allowed
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered

Endocrine therapy

* At least 4 weeks since prior endocrine therapy

  * Multiple lines of endocrine therapy for advanced disease allowed

Radiotherapy

* At least 4 weeks since prior radiotherapy and recovered

  * Prior radiotherapy for metastatic disease allowed

Surgery

* No prior major gastric surgery
* Prior surgery, including for metastatic disease, allowed

Other

* No other concurrent anticancer or investigational agents
* No concurrent antiretroviral therapy in HIV-positive patients
* Concurrent bisphosphonates allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-06; Primary Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Natasha Leighl, MD, FRCPC, Study Chair — Princess Margaret Hospital, Canada
Locations (4):
- Canada (4):
  - Margaret and Charles Juravinski Cancer Centre, Hamilton, Ontario
  - Cancer Care Ontario-London Regional Cancer Centre, London, Ontario
  - Ottawa Regional Cancer Centre, Ottawa, Ontario
  - Princess Margaret Hospital, Toronto, Ontario

REFERENCES:
- [Result] Leighl NB, Dent S, Clemons M, Vandenberg TA, Tozer R, Warr DG, Crump RM, Hedley D, Pond GR, Dancey JE, Moore MJ. A Phase 2 study of perifosine in advanced or metastatic breast cancer. Breast Cancer Res Treat. 2008 Mar;108(1):87-92. doi: 10.1007/s10549-007-9584-x. Epub 2007 Apr 26. PMID 17458693